CLINICAL TRIAL: NCT05664802
Title: e-HERO: Ending the HIV Epidemic in Rural Oklahoma
Acronym: e-HERO
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Northern Arizona University (Other)
Collaborators: Oklahoma State University (Other); Purdue University (Other); National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Principal Investigator, Julie Baldwin, Regents' Professor and Director, Northern Arizona University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: NAU IRB Protocol ID: 1827963-2; 3U54MD012388-05S2 (NIH)
Record Dates: First submitted 2022-12-16; First posted 2022-12-27 (Actual); Last update posted 2024-03-20 (Actual); Status verified 2024-03

CONDITIONS: Human Immunodeficiency Virus (HIV)
Keywords: Sexual and Gender Minorities; American Indian; HIV Testing
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Coitus

STUDY DESIGN:
Intervention Model Description: Centralized, computer-based group assignment using permuted blocks.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- e-HERO 2.0 (Experimental): The e-HERO intervention includes 10 modules, totaling approximately 2.5 hours of content. Across these modules, e-HERO uses diverse delivery methods to address HIV and STI knowledge, behavioral skills, HIV and STI testing intention, and instill self-efficacy to primary and secondary prevention behaviors. Those in the intervention condition will also engage in three virtual group discussion sessions with peer mentors.
  Interventions: Behavioral: e-HERO: Ending the HIV Epidemic in Rural Oklahoma
- e-HERO 1.0 (Active Comparator): e-HERO 1.0 contains the same number of modules as e-HERO. The control arm reflects HIV and STI information that is currently publicly available.
  Interventions: Behavioral: e-HERO: Ending the HIV Epidemic in Rural Oklahoma

INTERVENTIONS:
Behavioral: e-HERO: Ending the HIV Epidemic in Rural Oklahoma — A behavioral intervention utilizing online platforms to assess the impact of cultural tailoring of health education material.

SUMMARY:
The goal of this study is to increase HIV and syphilis testing and linkage to care, increase condom use, and promote PrEP uptake among sexual minority men (SMM) and American Indian (AI) men in rural Oklahoma, a state that is an Ending the HIV Epidemic (EHE) priority state. The proposed supplement aims to: refine our preliminary intervention strategy in partnership with a Community Advisory Board (CAB) and rural peer mentors, and to assess feasibility, acceptability, and preliminary impact of the e-HERO intervention.

DETAILED DESCRIPTION:
In the U.S., incidence rates of HIV and sexually transmitted infections (STIs) are disproportionately high among gay, bisexual, and other men who have sex with men-referred to herein as sexual minority men (SMM)-compared to men who have sex with women only. Similarly, rates of HIV infection have increased among American Indian (AI) men. This is a two-group, active-control RCT of the online e-HERO intervention. Participants (100 SMM; 100 AI men) will be randomized into two groups in equal proportions. This study evaluates two versions of an online sexual health intervention. The e-HERO intervention includes 10 modules, totaling approximately 2.5 hours of content. Across these modules, e-HERO uses diverse delivery methods (e.g., videos, interactive games) to address HIV and STI knowledge, behavioral skills, HIV and STI testing intention, and instill self-efficacy to primary and secondary prevention behaviors. Those in the intervention condition will also engage in three virtual group discussion sessions with peer mentors. The control condition contains the same number of modules as e-HERO. The control condition contains the same number of modules as e-HERO. The control arm reflects HIV and STI information that is currently available on many websites, with the aim to understand how the cultural tailoring of e-HERO modules improves upon information that is readily available online.

ELIGIBILITY:
Inclusion Criteria:

* Provide signed and dated informed consent form
* Be willing and able to follow study procedures and instructions and be available for the duration of the study
* Be between 17 and 29 years of age
* Be American Indian or a gay, bisexual, or other man who has sex with men. American Indian status is self-identified-no tribal enrollment verification will be required.
* Be a resident of Oklahoma, in a rural identified county

Exclusion Criteria:

* Anything that would place the individual at increased risk or preclude the individual's full compliance with, or completion of, the study.
* HIV diagnosis

Ages: 17 Years to 29 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes — Participants must identify as male, inclusive of transgender men.
Enrollment: 200 (Estimated)
Dates: Start 2022-12-01 (Actual); Primary Completion 2024-08-30 (Estimated); Study Completion 2024-08-30 (Estimated)

PRIMARY OUTCOMES:
HIV testing uptake | Assessed at the end of month 3 of the intervention.
  HIV testing uptake is assessed through the request of an at-home rapid HIV test through the e-HERO platforms.

SECONDARY OUTCOMES:
HIV testing intention | Baseline, 1 month, and 3 months
  Intention to get tested for HIV is assessed on a 6-point Likert scale (Extremely unlikely to get tested to Extremely likely to get tested).
STI testing intention | Baseline, 1 month, and 3 months
  Intention to get tested for STIs is assessed on a 6-point Likert scale (Extremely unlikely to get tested to Extremely likely to get tested).
PrEP consult with medical provider | 1 month and 3 months
  Single-item measure assessing if they have consulted with a medical provider among PrEP within the last month and/or 3 months.
Condom use | Baseline, 1 month, and 3 months
  Single-item assessment of condom use with sexual partner during the last sexual event.

CONTACTS AND LOCATIONS:
Overall Officials: Julie Baldwin, Ph.D., Principal Investigator — Northern Arizona University
Locations (1):
- Northern Arizona University, Flagstaff, Arizona, United States

IPD SHARING:
Plan to Share IPD: No